CLINICAL TRIAL: NCT05214352
Title: Using the Involvement Matrix for the Implication of Young People With Cerebral Palsy in the Elaboration of an Intervention Program to Encourage Participation in the Community.
Brief Title: Use of Involvement Matrix in Cerebral Palsy Into Spain and Brazil
Acronym: InMatrix-CP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Castilla-La Mancha (Other)
Responsible Party: Sponsor
Other Study IDs: Rpalomo02
Record Dates: First submitted 2021-12-05; First posted 2022-01-28 (Actual); Last update posted 2022-01-28 (Actual); Status verified 2022-01

CONDITIONS: Public and Patient Involvement; Patient Participation; Family Research; Participation
Keywords: family; research project; co-design
MeSH Terms: conditions — Patient Participation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- young population with cerebral palsy-Families-Therapist and researchers: The principal group is designed by all people who composed the research and who will work together in the intervention manual elaboration on the participation in the community.
  Interventions: Other: co-design in the intervention manual elaboration to increase the participation in the community

INTERVENTIONS:
Other: co-design in the intervention manual elaboration to increase the participation in the community — It will co-design an intervention manual between all participants (families, young people with cerebral palsy and therapists) and researchers, using the involvement matrix to increase the participation of young people in the community.
  Different focus grous will be created to work together and various online meetings, masterclass, workshops to increase the knowlodge in all groups.

SUMMARY:
Application of Involvement Matrix in young people with Cerebral Palsy (GMFCS levels IV and V) from 12 to 17 years old with the purpose of improving the participation of this group in community leisure activities

DETAILED DESCRIPTION:
The "Involvement Matrix" is a tool, which was built with organizations of patients, patients, parents, educators, doctors, and researchers, and supports the conversation and discussion about roles and expectations, aiming at authentic and sustainable alliances in research. It includes five participation roles: Listener, Co-thinker, Advisor, Partner and Decision-maker in three main phases of the research project: Preparation, Execution, and Implementation. The Involvement Matrix aims to be a guide for the project leader or researcher to dialogue with patients (public). Using the Matrix, agreements are made about the roles that the patient wishes to acquire and how they are involved in each phase. In this way, the empty cells in the Matrix are filled with specific activities.

Using the Involvement Matrix before and during the different phases of a project has the potential to help researchers and patients reach clear agreements about research and their participation. The tool can be used prospectively, to discuss the possible roles of patients in the different phases of the projects, and retrospectively to discuss whether the roles have been satisfactorily performed. It is known that some studies with PPI had children and young people with the most severe disabilities as active participants and with non-verbal communication, thus, the most effective ways to collaborate with this group should be developed and enhanced to encourage their involvement in research. Although periodicals on the PPI are increasing rapidly, a solid evidence base of the impact of the PPI on research is still lacking, as many publications relate to the PPI process in general and without addressing the real impact of the PPI on the research.

In this sense, the goal of this project is "to develop (co-production) an intervention program for young people with Cerebral Palsy (GMFCS levels IV and V) from 12 to 17 years old with the purpose of improving the participation of this group in community leisure activities and assess the viability of public involvement in the research project through the use of the Involvement Matrix ".

ELIGIBILITY:
Inclusion Criteria:

* young people diagnosed with Cerebral Palsy (CP) from 12 to 17 years old, levels IV-V within the Gross Motor Function Classification System (GMFCS)
* preserved cognitive status
* families willing to cooperate with the research, as well as the physiotherapists and occupational therapists that accept to participate in the study.

Exclusion Criteria:

* young people with an inadequate cognitive level (CI <70) to answer questions and collaborate, with other problems or diseases not associated with CP
* non-cooperative families, and physiotherapists and occupational therapists who do not agree to sign the informed consent form for inclusion in the study

Ages: 12 Years to 17 Years | Sex: All
Age Groups: Child
Study Population: The research will be carried out remotely (online) with 9 young people from 12 to 17 years old with cerebral palsy, GMFCS IV and V, their families and 6 healthcare professionals (physiotherapists and occupational therapists).
Sampling Method: Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2022-02-01 (Estimated); Primary Completion 2022-05-30 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
open questions and surveries | 12 weeks
  to obtain the experiences from young people with cerebral palsy, families and therapist.
  These questionnaires will be designed by patients and therapist to introduce the correct information
The PEM-CY: Participation and Environment Measure - Children and Youth | At baseline to know how is the participation in young people to increase it in the works groups.
  is a measure that evaluates participation in the home, at school, and in the community, alongside environmental factors within each of these settings.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Castilla-La Mancha, Toledo, Spain

IPD SHARING:
Plan to Share IPD: No
The protocol study will be shared with other researchers

REFERENCES:
- [Result] Mitchell SJ, Slowther AM, Coad J, Akhtar S, Hyde E, Khan D, Dale J. Ethics and patient and public involvement with children and young people. Arch Dis Child Educ Pract Ed. 2019 Aug;104(4):195-200. doi: 10.1136/archdischild-2017-313480. Epub 2018 Feb 9. PMID 29440127
- [Result] Alderson H, Brown R, Smart D, Lingam R, Dovey-Pearce G. 'You've come to children that are in care and given us the opportunity to get our voices heard': The journey of looked after children and researchers in developing a Patient and Public Involvement group. Health Expect. 2019 Aug;22(4):657-665. doi: 10.1111/hex.12904. Epub 2019 May 21. PMID 31115138
- [Result] Forsyth F, Saunders C, Elmer A, Badger S. 'A group of totally awesome people who do stuff' - a qualitative descriptive study of a children and young people's patient and public involvement endeavour. Res Involv Engagem. 2019 Mar 12;5:13. doi: 10.1186/s40900-019-0148-0. eCollection 2019. PMID 30915233
- [Result] Costello W, Dorris E. Laying the groundwork: Building relationships for public and patient involvement in pre-clinical paediatric research. Health Expect. 2020 Feb;23(1):96-105. doi: 10.1111/hex.12972. Epub 2019 Oct 18. PMID 31625656
- [Result] Boland L, Graham ID, Legare F, Lewis K, Jull J, Shephard A, Lawson ML, Davis A, Yameogo A, Stacey D. Barriers and facilitators of pediatric shared decision-making: a systematic review. Implement Sci. 2019 Jan 18;14(1):7. doi: 10.1186/s13012-018-0851-5. PMID 30658670
- [Result] Smits DW, van Meeteren K, Klem M, Alsem M, Ketelaar M. Designing a tool to support patient and public involvement in research projects: the Involvement Matrix. Res Involv Engagem. 2020 Jun 16;6:30. doi: 10.1186/s40900-020-00188-4. eCollection 2020. PMID 32550002
- [Result] van Schelven F, van der Meulen E, Kroeze N, Ketelaar M, Boeije H. Patient and public involvement of young people with a chronic condition: lessons learned and practical tips from a large participatory program. Res Involv Engagem. 2020 Sep 30;6:59. doi: 10.1186/s40900-020-00234-1. eCollection 2020. PMID 33005440